CLINICAL TRIAL: NCT02225990
Title: Implementation of Gait Coordination, Mobility, and Fitness Training for Enhanced Quality of Life and Participation in Life Roles
Brief Title: Implementation of Comprehensive Stroke Rehabilitation Therapy for Enhanced Quality of Life
Acronym: QualPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400568
Record Dates: First submitted 2014-08-15; First posted 2014-08-26 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: stroke; stroke rehabilitation; stroke therapy
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (4):
- Standard of Care, Sub-Acute (Active Comparator): This group will receive standard of care stroke rehabilitation therapy.
  Interventions: Other: Standard of Care, Sub-Acute
- Standard of Care, Chronic (Active Comparator): This group will receive standard of care stroke rehabilitation therapy.
  Interventions: Other: Standard of Care, Chronic
- Experimental Group, Sub-Acute (Experimental): This group consists of sub-acute stroke patients who are between three weeks and six months post-stroke and will receive the QualPro protocol. If the participant is an inpatient at Shands Rehabilitation Hospital at the beginning of the study, his/her first three weeks of research therapy sessions will take place at the Shands Rehabilitation Hospital. After being discharged, the remainder of the study sessions will take place at either UF Health Rehab Center- Magnolia Parke or in the North Tower (6th floor) physical therapy department of Shands Hospital.
  Interventions: Other: Experimental Group, Sub-Acute
- Experimental Group, Chronic (Experimental): This group consists of chronic stroke patients who are greater than six months post-stroke and will receive the QualPro protocol. The study sessions will take place at either UF Health Rehab Center-Magnolia Parke or in the North Tower (6th floor) physical therapy department of Shands Hospital.
  Interventions: Other: Experimental Group, Chronic

INTERVENTIONS:
Other: Experimental Group, Sub-Acute — For the sub-acute experimental group, the intervention schedule will be as follows: six months of individual therapy five times weekly (1 - 2.5 hours/session); 6 months of 'refresher' individual therapy twice monthly (1 - 2.5 hours/session) + group therapy up to three times weekly (1 hour/session); and 1 year of group therapy, up to three times weekly (1 hour/session) + 1 'refresher' individual therapy session every 3 months for a total study duration of 2 years.
  Arms: Experimental Group, Sub-Acute
Other: Experimental Group, Chronic — For the chronic experimental group, the intervention schedule will be as follows: six months of individual therapy five times weekly (1 - 2.5 hours/session); 6 months of 'refresher' individual therapy twice monthly (1 - 2.5 hours/session) + group therapy up to three times weekly (1 hour/session); and 1 year of group therapy, up to three times weekly (1 hour/session) + 1 'refresher' individual therapy session every 3 months for a total study duration of 2 years.
  Arms: Experimental Group, Chronic
Other: Standard of Care, Sub-Acute — This group will receive standard of care stroke rehabilitation therapy.
  Arms: Standard of Care, Sub-Acute
Other: Standard of Care, Chronic — This group will receive standard of care stroke rehabilitation therapy.
  Arms: Standard of Care, Chronic

SUMMARY:
The purpose of this research study is to implement into clinical practice, the comprehensive QualPro protocol for stroke survivors, which includes gait coordination, balance, mobility, and fitness training. Feasibility will be tested in the clinical environment by providing the intervention, measuring patient outcomes, and identifying the obstacles to insurance payment for the QualPro intervention. By productively addressing issues of implementation, the hypotheses of this study include proven feasibility in the clinical environment and clinically significant gains for stroke patients in the areas of strength, balance, gait coordination, endurance, physical function, and increased life role participation.

DETAILED DESCRIPTION:
This comprehensive intervention targets the impairments preventing recovery to normal and safe gait, mobility, function, and life role participation (quality of life). It has been tested in chronic stroke survivors and found efficacious.

The QualPro protocol will include three phases, all of which contain components previously mentioned. The QualPro protocol includes implementation of gait coordination training to address weakness, impaired endurance, and dyscoordination. The protocol will include implementation of balance training for falls prevention composed of Yang style, 24-posture, short-form Tai Chi. Additionally, the QualPro protocol will include implementation of aerobic training for fitness, health, and endurance of stroke survivors, which will be composed of low-volume, high intensity interval training (HIIT) on a cycle ergometer. Strength exercises will also be included. All exercises will address weakness, impaired endurance, and dyscoordination.

The long-range financial goal of this research study is to realize the cost savings of implementing the proposed combination of interventions that will preclude much of the very costly and downwardly spiraling sequellae currently observed after stroke, and that currently costs managed care and insurance companies an exorbitant and unnecessary amount of precious resources.

ELIGIBILITY:
Inclusion Criteria:

* Cognition sufficiently intact to give valid informed consent to participate.
* Sufficient endurance to participate in rehabilitation sessions.
* Ability to follow 2 stage commands.
* Medically stable
* Age > 21 years
* Impaired ambulation as follows: inability to flex the knee and ankle in the sagittal plane, in a normal manner so the foot clears the floor; inability to control normal knee angle during single limb weight bearing during stance phase.
* Trace contraction of hip, knee, and ankle flexors and extensors.
* Passive range of motion (ROM) at hip, knee, ankle greater than or equal to normal gait kinematics.
* Reported comfort of surface FES at a stimulus level producing a visible or palpable muscle contraction of ankle dorsiflexors.
* Greater than 3 weeks post-stroke.
* Living in the community and able to travel to training and assessment sites.
* Approval of participation by primary care physician

Exclusion Criteria:

* Acute or progressive cardiac, renal, respiratory, neurological disorders or malignancy.
* Active psychiatric diagnosis or psychological condition, or active drug/alcohol abuse.
* Lower motor neuron damage or radiculopathy.
* More than one stroke.
* Cerebellar dysfunction.
* Fugl-Meyer lower limb motor sub-score greater than 32.
* Severe obesity (body mass index > 35)
* For the chronic group: current participation in physical therapy or cardiopulmonary rehabilitation.
* Significant visual impairment affecting capability to gauge movement accuracy.
* Current enrollment in any clinical trial
* Planning to relocate out of the greater Gainesville, FL area during the study period
* Unable to communicate sufficiently with study personnel
* Clinical judgement regarding safety or non-compliance
* Refusal to be recorded by video for gait assessment

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Patient response to QualPro intervention in the clinical environment | 24 months
  Implementation of the comprehensive QualPro protocol into clinical practice will be done in order to determine patient outcomes during interventions of gait coordination, balance, mobility, and fitness training.

SECONDARY OUTCOMES:
Cost savings of implementation of the QualPro Protocol | 24 Months
  Information with respect to the cost of standard care and cost of the proposed care model will be collected and compiled in order to determine feasibility in the clinical environment.

CONTACTS AND LOCATIONS:
Overall Officials: Janis J. Daly, PhD, MS, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Health Rehab Center- Magnolia Parke, Gainesville, Florida
  - UF Health Shands Rehab Hospital, Gainesville, Florida
  - Brain Rehabilitation Research Center, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided